CLINICAL TRIAL: NCT05381116
Title: A Prospective, Sham-Controlled, Safety and Efficacy Study of a Smart, Self-Adjusting, Surgery-Free, Wearable Bladder Modulation and Digital Health System With Objective Confirmation of Nerve Activation for Use in Home by Subjects With Overactive Bladder Syndrome
Brief Title: A Sham-Controlled Study to Evaluate the Safety and Efficacy of a Smart, Self-Adjusting, Surgery-Free, Wearable Bladder Neuromodulation System for Overactive Bladder
Acronym: REDUCEOAB
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor Initiated
Sponsor: Avation Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AMHOAB2101
Record Dates: First submitted 2022-05-03; First posted 2022-05-19 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Overactive Bladder; Urinary Urge Incontinence; Urge Incontinence
Keywords: Overactive Bladder; OAB; Urinary Incontinence; Neuromodulation; Bioelectronic Medicine; Urologic Disorders; Wearable; Digital Health; Closed-Loop; EMG; Sham; Continuous Sensing; Automatic Adjustment
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge; Urinary Incontinence; Urologic Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Experimental Arm (Active Comparator): Avation System
  Interventions: Device: Avation System
- Control Arm (Sham Comparator): Sham Avation System
  Interventions: Device: Sham Avation System

INTERVENTIONS:
Device: Avation System — Subjects will perform therapy with active Avation System three (3) times a week for thirty (30) minutes each time over a 12-week period. At the end of the twelve (12) weeks of therapy, eligible Subjects from the Active Arm will be offered the opportunity to participate in the additional twenty one (21) month Open-Label Phase.
  Arms: Experimental Arm
Device: Sham Avation System — Subjects will perform therapy with sham Avation System three (3) times a week for thirty (30) minutes each time over a 12-week period. At the end of the twelve (12) weeks of therapy, all Subjects from the Sham Arm will be offered the opportunity to crossover and participate in the additional twenty one (21) month Open-Label Phase.
  Arms: Control Arm

SUMMARY:
This is a prospective, multi-center, sham-controlled study comparing the safety and effectiveness of the self-adjusting, surgery-free, wearable Active System to a Sham System on adult Subjects diagnosed with OAB.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female and 18 years of age or older at the time of enrollment
2. Willing and capable of giving informed consent
3. Willing and able to comply with all Study-related requirements and procedures
4. Have been diagnosed or have symptoms of OAB for at least 3 months prior to enrollment
5. Have an average of 11 or more voiding events and/or 3 or more incontinent events per 24-hour period in a 3-Day Bladder Diary(a minimum of 30 voiding events over the 3 days measured by the Diary)
6. If currently on medications that may affect their OAB symptoms, is on a stable dose (no new, discontinued, or change in dose) of all prescribed medications for at least 4 weeks prior to enrollment or throughout the Study
7. Female Subjects of child-bearing potential must have a negative urine dip stick pregnancy test at baseline

Exclusion Criteria:

1. Has been diagnosed with incontinence due to neurogenic bladder(stroke, CNS tumors, Parkinson's etc.)
2. Have failed a third line treatment (PTNS, Botox or SNS) for their OAB because of lack of effectiveness within the 2 years prior to enrollment
3. Have evidence of an uncontrolled active disruptive psychological or psychiatric disorder or other known condition significant enough to impact perception of pain, compliance of intervention and/or ability to evaluate treatment outcomes, in the opinion of the Investigator
4. Has or had a significant untreated substance use disorder or polysubstance use disorder stemming from dependency-producing medications, alcohol, and/or illicit drugs less than 6 months prior to enrollment
5. Are planning to or have scheduled a surgery, for any condition, that would require catheterization, or a prolonged hospital stay and affect the ability to ambulate, use the toilet, or complete Therapy during the first 12 weeks of the Study
6. Has symptoms of, been diagnosed, or being actively treated for benign prostatic hyperplasia or prostate cancer (weak stream, straining, hesitancy, or intermittency)
7. Have a pacemaker or implanted defibrillator
8. Has a neurological disorder that affects the bladder or a diagnosis of interstitial cystitis, radiation cystitis, or fistulas
9. Incontinence due to stress-predominant mixed urinary incontinence (greater that 60% of the time)or being actively treated for stress urinary incontinence(Diagnosed or by review of the Baseline 3-Day Bladder Diary)
10. Has been diagnosed with or has symptoms of polyuria (>2500 cc urine output per day)
11. Has urinary retention or incomplete bladder emptying
12. Have a documented current or reoccurring Urinary Tract Infection (3 or more in the months prior to enrollment)
13. Have had Botox treatment for their OAB in the previous 8 months
14. Have used TENS anywhere on the body within the last year for any reason or anticipated use of TENS within 12 weeks of enrollment in pelvic region, back or legs for any reason
15. Had PTNS treatment for OAB within 6 months prior to enrollment.
16. Use of investigational drug/device Therapy, for any reason, within past 12 weeks
17. Current use or implantation of an implanted device for treatment of their OAB or incontinence (including but not limited to sacral nerve stimulators)
18. Participation in another clinical Study during the term of the Study
19. Pregnant or planning to become pregnant during the Study. Female Subjects of childbearing potential who become pregnant during the Study will be withdrawn from the Study and will be asked to sign a separate pregnancy consent form to allow the Investigator and Sponsor to follow up on the Subject's pregnancy and outcome
20. Has scar tissue, metal, or another implant or a large tattoo that might interfere with Therapy
21. Has a neurological disorder that causes abnormal sensations in the lower leg (loss of sensation or allodynia)
22. Has a skin condition, for example allergic reaction, rash or open wounds, in the area of where the Therapy Garment will be placed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2022-04-14 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
The proportion of Subjects with a successful response | Blinded Lead-In Portion of Study,12 Weeks
  The proportion of Subjects with a successful response, where success is defined as:
  For enrolled Subjects that meet the inclusion criteria for average voids per day (frequency): a Subject that achieves a 50% or greater reduction, from baseline (Visit 1) to Week 12 (Visit 4), in average voids per day relative to an upper normal limit of an average of 8 voids per day, or
  For enrolled Subjects that meet the inclusion criteria for incontinence events per day: a Subject that achieves a 50% or greater reduction from baseline (Visit 1) to Week 12 (Visit 4) in average incontinence events (IE) per day.

SECONDARY OUTCOMES:
Quality of Life Endpoints: Questionnaires | Length of Study, 24 months
  Evaluation of the Subject Quality of Life questionnaires used throughout the duration of the trial.

OTHER OUTCOMES:
Open-Label Phase Endpoints | Length of Study, 24 months
  During the Open-Label Phase, efficacy endpoints for enrolled Subjects that meet the inclusion criteria for average voids per day (frequency): a Subject that achieves a 50% or greater reduction, from baseline (Visit 1) in average voids per day relative to an upper normal limit of an average of 8 voids per day, or for enrolled Subjects that meet the inclusion criteria for incontinence events per day: a Subject that achieves a 50% or greater reduction from baseline (Visit 1) to in average incontinence events (IE) per day, except that Subjects initially enrolled in the Sham Arm will convert to Active Therapy (3x per week for 12 weeks followed by at least 1x per week for the remainder of the Study) and endpoints will be measured against their baseline (Visit 1) diary.
  .

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Eclipse Clinical Research, Tucson, Arizona
  - Women's Health Institute, Oak Lawn, Illinois
  - Ochsner Medical Center, New Orleans, Louisiana
  - Regional Urology, Shreveport, Louisiana
  - Flourish Research, San Antonio, Texas
  - Tranquil Medical Rsearch, Webster, Texas